CLINICAL TRIAL: NCT04666090
Title: A Prospective, One-arm, Single-center, Phase Ⅱ Clinical Study of Carrelizumab Combined With Chemotherapy and Antiangiogenic Drugs in the Neoadjuvant Treatment of Resectable Esophageal Squamous Cell Carcinoma
Brief Title: Carrelizumab, Chemotherapy and Apatinib in the Neoadjuvant Treatment of Resectable Esophageal Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-795
Record Dates: First submitted 2020-12-03; First posted 2020-12-14 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Squamous Cell Carcinoma; Neoadjuvant Therapy
Keywords: Carrelizumab; Neoadjuvant Treatment; Esophageal Squamous Cell Carcinoma; Apatinib
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Esophagectomy; Sampling Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carillizumab (Experimental): Preoperative neoadjuvant therapy for 2-3 cycles. Radical surgery is performed 4-6 weeks after the last dose. Postoperative radiotherapy is determined according to the clinical situation and pathological stage of the patient.
  Carillizumab can be maintained for a maximum of 1 year. During the study, patients were be followed until disease progression, withdrawal of informed consent, loss of follow-up, or death.
  Interventions: Drug: Carillizumab; Procedure: Esophagectomy; Other: Samples

INTERVENTIONS:
Drug: Carillizumab — administration regimen: Carillizumab 200mg, IV, D1; Albumin paclitaxel 150mg/m2, D1; Nedaplatin 50 mg/m2, D1; Apatinib 250mg Po D2-4. Preoperative neoadjuvant therapy for 2-3 cycles, one cycle every 14 days.
  Other Names: Esophagectomy; Collecting samples from participant
Procedure: Esophagectomy — Laparoscopy combined with thoracoscope radical resection of esophageal carcinoma
Other: Samples — Blood, Tumour and Saliva will be Collected from participant. Fate of sample is Destruction after use

SUMMARY:
China with high incidence of esophageal cancer, the number of new cases and deaths account for about 50% of the world every year. In the past few decades, surgery, radiotherapy, chemotherapy and other treatments were continuously improved, however, the mortality of esophageal squamous cell carcinoma patients was not significantly decreased.

For patients with locally advanced esophageal cancer, direct surgery is not effective. It is difficult to achieve radical resection by surgery merely, and even if many patients receive surgery, they may eventually have tumor recurrence and poor survival rate. Therefore, it is necessary to explore effective perioperative neoadjuvant treatment to reduce the risk of postoperative recurrence and improve the postoperative survival rate of patients.

According to the reports, the expression of PD-L1 in esophageal cancer was about 41.4%. Therefore, PD-1/ PD-L1 immunocheckpoint inhibitor may become a new method for the treatment of esophageal cancer. Preliminary clinical results showed that immunotherapy combined with chemoradiotherapy provided a synergies antitumor effect. Multiple clinical results showed that Carrillizumab provided higher overall response rate for advanced esophageal cancer.

However, in patients with locally advanced esophageal cancer, the efficacy of Carrillizumab combined with chemotherapy and apatinib for sequential radical surgery is still unclear. The purpose of this study is to observe and evaluate the efficacy and safety of Carrillizumab combined with chemotherapy and antiangiogenic drugs in the neoadjuvant therapy of resectable esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
Esophageal cancer is a common malignant tumor of the digestive tract. Every year, there are about 400,000 new cases of esophageal cancer in the world and about 300,000 people dying of this disease. China with high incidence of esophageal cancer, the number of new cases and deaths account for about 50% of the world every year. In the past few decades, surgery, radiotherapy, chemotherapy and other treatments were continuously improved, however, the mortality of esophageal squamous cell carcinoma patients was not significantly decreased. Early local invasion, lymph node metastasis and distant metastasis are the main causes of poor prognosis for the patients with esophageal squamous cell carcinoma.

For patients with locally advanced esophageal cancer, direct surgery is not effective. It is difficult to achieve radical resection by surgery merely, and even if many patients receive surgery, they may eventually have tumor recurrence and poor survival rate. Therefore, it is necessary to explore effective perioperative neoadjuvant treatment to reduce the risk of postoperative recurrence and improve the postoperative survival rate of patients.

In recent years, PD-1 antibody is undoubtedly the most dazzling star in the field of tumor therapy. It shows excellent efficacy in of the different kind of tumors. According to the reports, the expression of PD-L1 in esophageal cancer was about 41.4% (Meta-analysis of 1350 Chinese and Japanese subjects showed that the over-expression of PD-L1 tended to decrease overall survival). Therefore, PD-1/ PD-L1 immunocheckpoint inhibitor may become a new method for the treatment of esophageal cancer. Preliminary clinical results showed that immunotherapy combined with chemoradiotherapy provided a synergies antitumor effect. Multiple clinical results showed that Carrillizumab provided higher overall response rate for advanced esophageal cancer. It also provided superior progression free survival and overall survival compared with Pembrolizuma and paclitaxel. 2020 Chinese Society Of Clinical Oncology esophagus cancer guidelines recommended Carrillizumab as the first level for squamous cell carcinomas.

However, in patients with locally advanced esophageal cancer, the efficacy of Carrillizumab combined with chemotherapy and apatinib for sequential radical surgery is still unclear. The purpose of this study is to observe and evaluate the efficacy and safety of Carrillizumab combined with chemotherapy and antiangiogenic drugs in the neoadjuvant therapy of resectable esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. signed informed consent;
2. patients age 18 to 75 years old
3. primary resectable, histologically confirmed esophageal squamous cell cancer;
4. Esophageal squamous cell carcinoma the clinical stage was IIA-IVA (according to AJCC TNM stage, 8th edition).
5. ECOG PS 0-1.
6. No distant metastasis, the diseases could be resectable assessed by thoracic oncologist;

Exclusion Criteria:

1. with significant cardiovascular disease;
2. current treatment with anti-viral therapy or HBV;
3. Female patients who are pregnant or lactating;
4. history of malignancy within 5 years prior to screening;
5. active or history of autoimmune disease or immune deficiency;
6. signs of distant metastases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (PCR) | 1 month after surgery
  No residual invasive tumor cells were found in the pathological examination of resected specimens.

SECONDARY OUTCOMES:
Major Pathological Response (MPR) | 1 month after surgery
  In the pathological examination of resected specimens, the proportion of residual tumor cells was less than 10%.
Objective Response Rate (ORR) | 1 month after surgery
  The proportion of subjects with imaging PR or CR assessed according to RECIST 1.1 criteria
2-year and 5-year overall survival | 2-year and 5-year after surgery
  The proportion of all study cases in which no death from any cause occurred within 2 years and 5 years after surgery
2-year and 5-year disease-free survival | 2-year and 5-year after surgery
  No recurrence, distant metastasis, or death within 2 years and 5 years after surgery accounted for the proportion of all cases studied.
Incidence of Treatment-related Adverse Events | 1 month after surgery
  Incidence of Treatment-related Adverse Events as Assessed by CTCAE v5.0
R0 resection rate | 1 month after surgery
  The pathological results showed that the incision margin was negative and no residual cancer cells were found under the microscope
The changes in the peripheral blood immunoprofile among non-PCR (NPCR) and PCR patients | 3 month after surgery
  By using mass spectrometry (CyTOF) and bioinformatics pipelines, we comprehensively characterized the immune landscape in the peripheral blood of ESCC patients before and after anti-PD-1 immunotherapy, aiming to explore the immune subsets correlated with neoadjuvant immunotherapy response

CONTACTS AND LOCATIONS:
Overall Officials: Weilin Wang, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, China, China

REFERENCES:
- [Derived] Wu Z, Wu C, Zhao J, Wu C, Peng H, Wang Q, Bai R, Fang X, He H, Shen H, Wu M. Camrelizumab, chemotherapy and apatinib in the neoadjuvant treatment of resectable oesophageal squamous cell carcinoma: a single-arm phase 2 trial. EClinicalMedicine. 2024 Apr 6;71:102579. doi: 10.1016/j.eclinm.2024.102579. eCollection 2024 May. PMID 38618203